CLINICAL TRIAL: NCT04224207
Title: Management of Retinitis Pigmentosa by Wharton's Jelly Derived Mesenchymal Stem Cells: Preliminary Clinical Results
Brief Title: Management of Retinitis Pigmentosa by Mesenchymal Stem Cells by Wharton's Jelly Derived Mesenchymal Stem Cells
Acronym: WJ-MSC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01.11.2018/01
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Retinitis Pigmentosa; Inherited Retinal Dystrophy
Keywords: Retinitis pigmentosa; Wharton's jelly derived mesenchimal stem cell; Subtenon space; Umbilical cord
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Prospective, open-label clinical trial; The statistical comparisons were made primarily between the baseline and final values from the same eye. The parametric results for visual functions and structural changes were analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before application (Active Comparator): RP patients with progressive visual acuity and visual field loss: before stem cell application.
  Interventions: Biological: Wharton's jelly derived mesenchymal stem cell
- After application (Active Comparator): RP patients, after stem cell applications.
  Interventions: Biological: Wharton's jelly derived mesenchymal stem cell

INTERVENTIONS:
Biological: Wharton's jelly derived mesenchymal stem cell — The mesenchymal cells that were used in this study were isolated from Wharton's jelly of the umbilical cord that was collected allogenicly from a single donor with the mother's consent. All cell preparation and cultivation procedures were conducted in a current Good Manufacturing Practice (cGMP) accredited laboratory (Onkim Stem Cell Technologies, Turkey).Cells were solubilized from cryopreservation before being made ready for injection. Average cell viability for each treatment was over 90.0% and each patient received cell numbers between 2-6x106 in a 1.5 ml saline solution .

SUMMARY:
The aim of this study is to determine if umbilical cord Wharton's jelly derived mesenchymal stem cells implanted in sub-tenon space have beneficial effects on visual functions in retinitis pigmentosa patients by reactivating the degenerated photoreceptors in dormant phase.

DETAILED DESCRIPTION:
The retinal pigment epithelium (RPE) forms the outer blood-retinal barrier between photoreceptor cells and choroidal blood vessels. Photoreceptor cells are vitally and functionally dependent on the RPE. The conversion of blood glucose to ATP, synthesis of proteins in the visual cycle and removal of metabolic waste takes place in the RPE. For these important processes, various peptide growth factors and their receptors are synthesized in the RPE. More than 260 genes in the RPE are responsible for the production of these peptide fragments. Mutations in any of these genes as well as ischemic, physical or chemical RPE damage causes retinal degeneration. Retinal degeneration may be inherited, such as in retinitis pigmentosa (RP), Stargardt's disease, choroideremia, Best vitelliform dystrophy and Bietti's crystalline dystrophy. Retinal degeneration may also be acquired through genetic mechanisms, such as age-releated macular degeneration. In retinal degeneration, there is a developing loss of RPE and photoreceptors, regardless of the underlying cause.

Umbilical cord Wharton's jelly derived mesenchymal stem cells (WJ-MSCs) have significant paracrine and immunomodulatory properties. WJ-MSCs secrete trophic factors that stimulate RPE or secrete trophic factors that are similar to those produced by RPE. In studies using animal models, WJ-MSCs have been found to be effective in stopping the progression of retinal degeneration and for rescuing photoreceptors in the dormant phase. WJ-MSCs are hypoimmunogenic and have significant immunomodulatory properties. WJ-MSCs have been shown to suppress chronic inflammation and prevent apoptosis in animal models of neurodegenerative and ischemic retinal disorders. WJ-MSCs also stimulate progenitor cells in the retina and elicit self-repair mechanisms.

The aim of this preliminary clinical study is to investigate the efﬁcacy of deep sub-tenon injected WJ-MSCs as a stem cell treatment modality for the management of retinitis pigmentosa, which creates outer retinal degeneration. These functional and structural effects were investigated using microperimetry, electrophysiology and spectral domain optical coherence tomography (SD-OCT). To the best of our knowledge, this is the first prospective clinical study that utilizes a large number of RP cases, and cases that are in phase-3.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older;

  * Diagnosis of any phenotypic or genotypic variation of RP, confirmed by clinical history, fundus appearance, visual field (VF), electroretinogram (ERG) and genetic mutation analysis;
  * Having experienced various degrees of VF loss;
  * BCVA from 50 letters to 110 letters in the ETDRS chart testing (Topcon CC-100 XP, Japan);
  * Mean deviation (MD) values ranging between -33.0 and -5.0 dB with Compass visual field analysis (threshold 24-2, Sita Standard, Stimulus 3-white);
  * Intraocular pressure (IOP) of <22 mmHg.

Exclusion Criteria:

* • The presence of cataracts or other media opacity that might affect the VF, MD, or ERG recordings;

  * The presence of glaucoma, which causes visual field and optic disc changes;
  * The presence of any systemic disorder (e.g.,diabetes, neurological disease, or uncontrolled systemic hypertension) that may affect visual function;
  * The habit of smoking.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
ETDRS visual acuity | Change from baseline visual acuity at 6 months
  The visual acuity scores obtained from the baseline testing and the final examination were analyzed and compared statistically to determine effectiveness.

SECONDARY OUTCOMES:
Outer retinal thickness | Change from baseline outer retinal thickness at 6 months
  This is the thickness from the outer plexiform layer to the Bruch membrane in the 3x3 mm area of the fovea measured (and recorded automatically) by the multimodal imaging OCTA device.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University Biotechnology Institute, Ankara, Türkiye
  - Umut Arslan, Ankara, Türkiye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Musial-Wysocka A, Kot M, Sulkowski M, Badyra B, Majka M. Molecular and Functional Verification of Wharton's Jelly Mesenchymal Stem Cells (WJ-MSCs) Pluripotency. Int J Mol Sci. 2019 Apr 12;20(8):1807. doi: 10.3390/ijms20081807. PMID 31013696
- [Result] Leow SN, Luu CD, Hairul Nizam MH, Mok PL, Ruhaslizan R, Wong HS, Wan Abdul Halim WH, Ng MH, Ruszymah BH, Chowdhury SR, Bastion ML, Then KY. Safety and Efficacy of Human Wharton's Jelly-Derived Mesenchymal Stem Cells Therapy for Retinal Degeneration. PLoS One. 2015 Jun 24;10(6):e0128973. doi: 10.1371/journal.pone.0128973. eCollection 2015. PMID 26107378
- [Result] Rani S, Ryan AE, Griffin MD, Ritter T. Mesenchymal Stem Cell-derived Extracellular Vesicles: Toward Cell-free Therapeutic Applications. Mol Ther. 2015 May;23(5):812-823. doi: 10.1038/mt.2015.44. Epub 2015 Mar 19. PMID 25868399
- [Result] Canto-Soler V, Flores-Bellver M, Vergara MN. Stem Cell Sources and Their Potential for the Treatment of Retinal Degenerations. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(5):ORSFd1-9. doi: 10.1167/iovs.16-19127. PMID 27116661
- [Result] Garg A, Yang J, Lee W, Tsang SH. Stem Cell Therapies in Retinal Disorders. Cells. 2017 Feb 2;6(1):4. doi: 10.3390/cells6010004. PMID 28157165
- [Result] Mohamed EM, Abdelrahman SA, Hussein S, Shalaby SM, Mosaad H, Awad AM. Effect of human umbilical cord blood mesenchymal stem cells administered by intravenous or intravitreal routes on cryo-induced retinal injury. IUBMB Life. 2017 Mar;69(3):188-201. doi: 10.1002/iub.1608. Epub 2017 Feb 5. PMID 28164440
- [Result] Limoli PG, Vingolo EM, Limoli C, Scalinci SZ, Nebbioso M. Regenerative Therapy by Suprachoroidal Cell Autograft in Dry Age-related Macular Degeneration: Preliminary In Vivo Report. J Vis Exp. 2018 Feb 12;(132):56469. doi: 10.3791/56469. PMID 29553543
- [Derived] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly-derived mesenchymal stem cells: prospective analysis of 1-year results. Stem Cell Res Ther. 2020 Aug 12;11(1):353. doi: 10.1186/s13287-020-01870-w. PMID 32787913